CLINICAL TRIAL: NCT04734652
Title: A Phase 2b Study to Evaluate the Efficacy, Safety and PK of a Combination of Bictegravir, Emtricitabine, and Tenofovir Alafenamide Fumarate for Treatment of HIV-1 Infection in Patients With Drug Susceptible-TB on a Rifampicin-based Regimen
Brief Title: INSTI's For The Management of HIV-associated TB
Acronym: INSIGHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Collaborators: Johns Hopkins University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Cape Town (Other); Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Anushka Naidoo, Principal Investigator, Centre for the AIDS Programme of Research in South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPRISA 093; 1R01AI152142-01 (NIH)
Record Dates: First submitted 2021-01-11; First posted 2021-02-02 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: HIV/AIDS; Tuberculosis, Pulmonary
Keywords: Biktarvy® is a fixed dose combination; TLD- fixed-drug combination single tablet; Dolutegravir 50mg; HIV/AIDS; Tuberculosis, Pulmonary
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis, Pulmonary | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; dolutegravir; Lamivudine; Tenofovir

STUDY DESIGN:
Intervention Model Description: 80 participants for the Intervention Arm ART regimen which is a fixed-drug combination of a single tablet co-formulated regimen containing Bictegravir 50mg Emtricitabine 200mg and tenofovir alafenamide 25mg (BIC/FTC/TAF; Biktarvy®) that will be taken twice a day during rifampicin-containing TB treatment and 2 weeks after stopping TB treatment, thereafter the BIC/FTC/TAF single tablet co-formulation will be taken once daily.
  40 participants in the Control ARM: Dolutegravir 50mg /Lamivudine 300mg/ Tenofovir 300mg (TLD- fixed-drug combination single tablet) plus Dolutegravir 50mg evening dose during TB treatment and for two weeks after completion of TB treatment, then TLD once daily thereafter- as per Standard of Care (SOC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIC arm (Experimental): The Intervention Arm ART regimen is a fixed-drug combination of a single tablet co-formulated regimen containing Bictegravir 50mg Emtricitabine 200mg and tenofovir alafenamide 25mg (BIC/FTC/TAF; Biktarvy®) that will be taken twice a day during rifampicin-containing TB treatment and 2 weeks after stopping TB treatment, thereafter the BIC/FTC/TAF single tablet co-formulation will be taken once daily.
  Interventions: Combination Product: Biktarvy®
- DTG Arm (Active Comparator): Dolutegravir 50mg /Lamivudine 300mg/ Tenofovir 300mg (TLD- fixed-drug combination single tablet) plus Dolutegravir 50mg evening dose during TB treatment and for two weeks after completion of TB treatment, then TLD once daily thereafter- as per Standard of Care (SOC)
  Interventions: Combination Product: TLD- fixed-drug combination single tablet

INTERVENTIONS:
Combination Product: Biktarvy® — Biktarvy® is a fixed dose combination, single tablet containing bictegravir (BIC), emtricitabine (FTC), and tenofovir alafenamide (TAF) for oral administration.
  BIC is an integrase strand transfer inhibitor (INSTI). FTC, a synthetic nucleoside analog of cytidine, is an HIV nucleoside analog reverse transcriptase inhibitor (HIV NRTI). TAF, an HIV NRTI, is converted in vivo to tenofovir, an acyclic nucleoside phosphonate (nucleotide) analog of adenosine 5'-monophosphate. Each tablet contains 50 mg of BIC (equivalent to 52.5 mg of bictegravir sodium), 200 mg of FTC, and 25 mg of TAF (equivalent to 28 mg of tenofovir alafenamide fumarate) and the following inactive ingredients: croscarmellose sodium, magnesium stearate, and microcrystalline cellulose.
  Arms: BIC arm
Combination Product: TLD- fixed-drug combination single tablet — Standard of care Dolutegravir-based regimen
  Other Names: Dolutegravir 50mg /Lamivudine 300mg/ Tenofovir 300mg
  Arms: DTG Arm

SUMMARY:
This study is being conducted to assess the antiretroviral activity of a fixed-drug, single tablet, combination of Bictegravir 50mg/ Emtricitabine 200mg/ Tenofovir alafenamide 25mg (Biktarvy®) dosed twice daily in HIV-1 infected, ART-naïve patients with TB co-infection receiving a rifampicin-based tuberculosis (TB) treatment regimen. This study will assess the activity of Bictegravir and dolutegravir-containing ART regimens in patients with drug-susceptible TB through 48 weeks

DETAILED DESCRIPTION:
Primary objective: To characterize viral suppression rates (proportion of patients with suppressed viral load) at week 24 in the BIC arm

Secondary objectives:

To characterize viral suppression rates at weeks 12, 24 and 48 in the standard of care treatment (SOC) arm (currently, TDF 300mg/3TC 300mg/DTG 50mg) and at weeks 12 and 48 in the BIC/FTC/TAF arm.

To compare the pharmacokinetics (PK) of BIC when given twice daily and co-administered with Rifampicin during tuberculosis treatment vs when given alone after discontinuation of Rifampicin

To assess the incidence of TB associated IRIS in each arm, through week 24.

To characterize the tolerability of treatment in each arm by assessing frequency of clinician-initiated treatment interruptions or switches through week 48.

To assess frequency of ART drug resistance mutations in participants with detectable viral load at study visit weeks 24 and 48.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age with Karnofsky score ≥ 70
* Confirmed rifampicin-susceptible tuberculosis and/or
* On first-line rifampicin-based tuberculosis treatment (not > 8 weeks at the time of enrolment)
* Documented HIV-1 infection, ART-naïve OR ART non-naïve (patients to have no exposure to ART medication at least ≥ 3 months at the time of enrollment)
* Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73m2
* Alanine aminotransferase (ALT) ≤3 times the upper limit of normal (ULN)
* Total bilirubin ≤2.5 times ULN
* Creatinine ≤2 times ULN
* Hemoglobin ≥ 7.0 g/dL (6.5 g/dL for females)
* Platelet count ≥ 50,000/mm3
* Absolute Neutrophil Count (ANC) ≥650/mm3
* Able and willing to provide written informed consent
* Female patients agree to use both a barrier and a non-barrier form of contraception during the study, starting at least 14 days prior to enrolment

Exclusion Criteria:

* Pregnancy or breastfeeding (or planned pregnancy within 12 months of study entry)
* Prior use of antiretroviral drugs for pre-exposure prophylaxis (PrEP) or post-exposure prophylaxis (PEP) < 3 months at the time of enrolment
* Hepatitis B surface antigen positive OR Hepatitis B virus (HBV) infection OR active systemic infections (other than HIV-1 infection) requiring systemic antibiotic or antifungal therapy current or within 30 days prior to baseline that could, in the opinion of the investigator, interfere with study procedures or assessment of study outcomes
* Participants with a CD4+ cell count of < 50 cells/ μl
* Any verified Grade 4 laboratory abnormality, with the exception of, Grade 4 triglycerides. A single repeat test is allowed during the Screening period to verify a result
* Patients on metformin (> 500mg, 12hourly)
* Patients with an uncontrolled psychiatric co-morbidity. Patients who, in the investigator's judgment, pose a significant suicidality risk. Recent history of suicidal behavior and/or suicidal ideation may be considered as evidence of serious suicide risk
* Other condition or circumstance deemed by clinician/investigators to be detrimental to patient safety or study conduct
* Unwilling to be part of the main pharmacokinetic (PK) study and have PK blood draws done (NB there is a semi-intensive PK substudy which is optional)

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anushka Naidoo, PhD, Principal Investigator — Centre for the AIDS Programme of Research in South Africa (CAPRISA); Kelly Dooley, MD, Principal Investigator — Vanderbilt University Medical Center; Kogieleum Naidoo, PhD, Study Director — Centre for the AIDS Programme of Research in South Africa
Locations (1):
- CAPRISA Springfield Clinical Research Site, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data generated under this project will be shared in accordance with CAPRISA, and NIH-SAMRC policies, including the NIH Data Sharing Policy. Research data that documents, supports, and validates research findings will be made available after the main findings from the final research data set have been accepted for publication.
Supporting Information: Study Protocol
Time Frame: Not longer than 12 months after first publication of results. In accordance with WHO stipulations, summary results or a link to summary results will be reported within the trial registration record within 12 months of the study completion date.
Access Criteria: Access to databases and associated software tools generated under the project will be available for educational, research, and non-profit purposes from bona-fide researchers and/or research organisations.

REFERENCES:
- [Derived] Naidoo A, Naidoo K, Letsoalo MP, Wasmann RE, Dorse G, Perumal R, Moosa MS, Osuala EC, Boodhram R, Chimukangara B, Wiesner L, Israelski D, Denti P, Rooney JF, Dooley KE; INSIGHT Study Team. Fixed-dose combination bictegravir-emtricitabine-tenofovir alafenamide twice-daily for treatment of HIV during rifampicin-based tuberculosis treatment (INSIGHT Study): a phase 2b, open-label, randomised non-comparative trial. Lancet HIV. 2026 Jan;13(1):e9-e20. doi: 10.1016/S2352-3018(25)00200-0. Epub 2025 Dec 1. PMID 41344350
- [Derived] Naidoo A, Dooley KE, Naidoo K, Padayatchi N, Yende-Zuma N, Perumal R, Dorse G, Boodhram R, Osuala EC. INSTIs for the management of HIV-associated TB (INSIGHT study): a phase 2b study to evaluate the efficacy, safety and pharmacokinetics of a combination of bictegravir, emtricitabine and tenofovir alafenamide fumarate for the treatment of HIV-1 infection in patients with drug-susceptible tuberculosis on a rifampicin-based treatment regimen: a phase 2b open-label randomised controlled trial. BMJ Open. 2022 Nov 10;12(11):e067765. doi: 10.1136/bmjopen-2022-067765. PMID 36356989

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential study participants were recruited from pre-approved clinics and hospitals. A pre-screening checklist was utilized by the Recruiters to select potential study participants.
Period: Overall Study
Arm/Group | BIC Arm | DTG Arm
Started | 80 | 42
Completed | 78 | 41
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIC Arm | DTG Arm | Total
Number analyzed (Participants) | 80 | 42 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 42 | 122
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 43
  Male | 55 | 24 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 80 | 42 | 122
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 80 | 42 | 122
Age, median range [Median (Full Range); unit: years] | 35 [19 to 56] | 35 [22 to 60] | 35 [19 to 60]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Viral Suppression at Week 24
Description: Viral suppression rate (HIV-1 RNA <50 copies/mL) at week 24 in the BIC arm (using the FDA snapshot algorithm).
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | BIC Arm | DTG Arm
Number analyzed (Participants) | 80 | 42
Participants
  Efficacy in PWH & TB through Week 24 ITT population | 75 | 40
  Treatment failure | 0 | 0

2. Secondary Outcome: Viral Suppression Rates (HIV-1 RNA <50 Copies/mL) at Weeks 12, 24 and 48 in the DTG Arm and at 12 and 48 Weeks in the BIC Arm
Description: To characterize viral suppression rates at weeks 12, 24 and 48 in the standard of care treatment (SOC) arm (currently, TDF 300mg/3TC 300mg/DTG 50mg) and at weeks 12 and 48 in the BIC/FTC/TAF arm.
Time Frame: Week 12 and 48
Reporting Status: Not Posted

3. Secondary Outcome: BIC Drug Concentrations ("Area Under the Plasma Concentration Versus Time Curve (AUC)"
Description: To assess BIC drug levels (AUC) when given twice daily and co-administered with Rifampicin vs. during TB treatment vs when given alone after TB treatment completion
Time Frame: Week 4, 8, 12, 24,32 and 40
Reporting Status: Not Posted

4. Secondary Outcome: BIC Drug Concentrations [Peak Plasma Concentration (Cmax)]
Description: To assess BIC drug levels (Cmax) when given twice daily and co-administered with Rifampicin vs. during TB treatment vs when given alone after TB treatment completion
Time Frame: Week 4, 8, 12, 24, 32 and 40
Reporting Status: Not Posted

5. Secondary Outcome: BIC Drug Concentrations [Trough/Minimum Plasma Concentration Ctrough)
Description: To assess BIC drug levels ( Ctrough) when given twice daily and co-administered with Rifampicin vs. during TB treatment vs when given alone after TB treatment completion
Time Frame: Week 4, 8 12, 24, 32 and 40
Reporting Status: Not Posted

6. Secondary Outcome: The Incidence of TB Associated IRIS
Description: To assess the incidence of TB associated IRIS in each arm
Time Frame: Through week 24
Reporting Status: Not Posted

7. Secondary Outcome: The Tolerability of Treatment in Each Arm
Description: To characterize the tolerability of treatment in each arm by assessing frequency of clinician-initiated treatment interruptions or switches through week 48
Time Frame: Through week 48
Reporting Status: Not Posted

8. Secondary Outcome: Frequency of ART Drug Resistance Mutations in Participants With Detectable Viral Load at Weeks 24 and 48
Description: To assess frequency of ART drug resistance mutations in participants with detectable viral load at weeks 24 and 48
Time Frame: Week 24 and 48.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 48 weeks
Description: Adverse events defined as DAIDS Toxicity Table
Arm/Group | BIC Arm | DTG Arm
All-Cause Mortality (participants affected / at risk) | 0/80 | 1/42
Serious Adverse Events (participants affected / at risk) | 11/80 | 3/42
Other Adverse Events (participants affected / at risk) | 0/80 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIC Arm (N=80) | DTG Arm (N=42)
Death (General disorders) | 0 (0) | 1 (1) — Hemoptysis, Grade 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Dyspnea Pneumonia Pyrexia IRIS associated TB
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Gastritis Vomiting Haematemesis
Shortness of breath (Infections and infestations) | 1 (1) | 0 (0) — Community acquired pneumonia Rash NOS
Cardiac failure investigations (Cardiac disorders) | 1 (1) | 0 (0) — cardiac failures
Left facial weakness and unsteady gait (Infections and infestations) | 1 (1) | 0 (0) — Tuberculosis of mastoid
Invasive fungal disease of ear. Chronic lung disease (Infections and infestations) | 1 (1) | 0 (0) — Ear infection fungal
Attempted suicide (Psychiatric disorders) | 1 (1) | 0 (0) — Parasuicide
Severe anaemia and renal impairment (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Anaemia
Investigation of left-sided weakness (Nervous system disorders) | 1 (1) | 0 (0) — Cerebrovascular accident NOS
Possible septic right hip (possible IRIS TB or infective aetiology) (Infections and infestations) | 1 (1) | 0 (0) — Cellulitis
Elevated conjugated hyperbilirubinemia (Investigations) | 1 (1) | 0 (0) — Conjugated bilirubin level increased
Underlying lung pathology with left upper zone nodules post completion of TB treatment# (Infections and infestations) | 1 (1) | 0 (0) — Klebsiella pneumoniae pneumonia Pneumocystis jirovecii pneumonia
New onset generalized tonic-clonic seizures (Nervous system disorders) | 1 (1) | 0 (0) — Seizures
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Ankle fracture
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — Miscarriage of pregnancy
Left lower leg cellulitis (Vascular disorders) | 0 (0) | 1 (1) — DVT

LIMITATIONS AND CAVEATS:
Non-comparative design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT04734652/Prot_001.pdf
  • Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT04734652/SAP_003.pdf
  • Informed Consent Form (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT04734652/ICF_002.pdf